CLINICAL TRIAL: NCT00323765
Title: Plasticity in Cervical Dystonia
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060157; 06-N-0157
Record Dates: First submitted 2006-05-09; First posted 2006-05-10 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-05-20

CONDITIONS: Cervical Dystonia
Keywords: Transcranial Magnetic Stimulation (TMS); Cervical Dystonia; Plasticity; Healthy Volunteer; HV
MeSH Terms: conditions — Torticollis

SUMMARY:
This study will identify changes that occur in the part of the brain that controls hand movements in patients with cervical (neck) dystonia. Patients with dystonia have muscle spasms that cause abnormal postures while trying to perform a movement. In focal dystonia, just one part of the body, such as the hand, neck or face, is involved. The study will compare findings in healthy volunteers and patients with cervical dystonia to learn more about the condition.

Healthy volunteers and patients with cervical dystonia 18 years of age and older may be eligible to participate. Candidates are screened with a medical history and physical examination. Participants undergo the following tests:

Somatosensory evoked potentials (Visits 1 and 2)

This test examines how sensory information travels from the nerves to the spinal cord and brain. An electrode placed on an arm or leg delivers a small electrical stimulus and additional electrodes placed on the scalp, neck and over the collarbone record how the impulse from the stimulus travels over the nerve pathways.

Transcranial Magnetic Stimulation (Visits 2, 3 and 4)

This procedure maps brain function. A wire coil is held on the scalp. A brief electrical current passes through the coil, creating a magnetic pulse that stimulates the brain. The stimulation may cause a twitch in muscles of the face, arm, or leg, and the subject may hear a click and feel a pulling sensation on the skin under the coil.

Nerve conduction studies (Visits 2, 3 and 4)

This test measures how fast nerves conduct electrical impulses and the strength of the connection between the nerve and the muscle. Nerves are stimulated through small wire electrodes attached to the skin and the response is recorded and analyzed.

Surface electromyography (Visits 2, 3 and 4)

Electrodes are placed on the front and back of the neck muscles to measure the electrical activity of the muscles.

DETAILED DESCRIPTION:
Objectives

The main objective of this proposal is to evaluate plasticity in patients with cervical dystonia. Neither abnormal Hebbian nor non-Hebbian plasticity has been studied for cervical dystonia.

Our specific objectives are to show that:

1. In patients with cervical dystonia, Hebbian plasticity can be induced by using paired associative stimulation (PAS) of the dystonic sternocleidomastoid muscle (SCM) muscle and will be enhanced compared to that of healthy subjects.
2. In patients with cervical dystonia, non-Hebbian plasticity can be induced by using transcutaneous electrical nerve stimulation (TENS) of the dystonic SCM muscle and will be enhanced compared to that of healthy subjects.
3. In patients with cervical dystonia, Hebbian and non-Hebbian plasticity can be induced by dual stimulation (DS) of the dystonic SCM muscle, this effect will be greater than PAS or TENS alone, and it will be enhanced compared to that of healthy subjects.

Study Population

We will study 22 patients with cervical dystonia and 22 healthy subjects for a total of 44 subjects.

Study Design

Subjects will participate in 4 different sessions:

Visit 1: clinical screening (1 hour) and sensory evoked potential (SEP) assessment (2 hours, total of 3 hours).

Visit 2: PAS session of the target muscle and monitoring of cortical excitability before (T0), immediately after (T1), 45 minutes after (T2) and 90 minutes after T(3) (Total of 4 hours).

Visit 3: TENS session of the target muscle and monitoring of cortical excitability before (T0), immediately after (T1), 45 minutes after (T2) and 90 minutes after T(3) (Total of 4 hours).

Visit 4: DS session of the target and monitoring of cortical excitability before (T0), immediately after (T1), 45 minutes after (T2) and 90 minutes after T(3) (Total of 4 hours).

Outcome Measures

The electrophysiological effects of the interventions will be assessed by the size of motor evoked potentials (MEP), resting and active motor threshold (RMT and AMT), and a transcranial magnetic stimulation (TMS) input-output curve. The activity of intracortical interneurons mediating long intracortical inhibition (LICI) will be assessed by paired-pulse TMS. The effect of afferent input on intracortical processes (long afferent inhibition, LAI) will be assessed by stimulating the skin overlying the sternocleidomastoid muscle (SCM).

ELIGIBILITY:
* INCLUSION CRITERIA:
* Healthy volunteers (aged 18 or older) who are willing to participate
* Patients (aged 18 and older) with idiopathic cervical dystonia that show a clear asymmetric involvement of the SCM muscles with lateral rotation of the head in the coronal or longitudinal plane

EXCLUSION CRITERIA:

* Subjects with additional significant neurological disorder, current use or a history of alcohol or drug abuse, psychiatric disorder requiring hospitalization or prolonged treatment such as substance abuse addiction, head injury with loss of consciousness, epilepsy.
* Subjects with significant hearing loss
* Subjects receiving drugs with significant action on the central nervous system
* Subjects who have been treated with botulinum toxin injections less than 3 months prior to their participation in the study
* Subjects who are taking any oral medication for dystonia at the time of the study

The following exclusion criteria are due to the use of transcranial magnetic stimulation:

* Subjects with cardiac pacemakers, implanted medication pumps
* Subjects with eye, blood vessel, cochlear, or eye implants
* Subjects with increased intracranial pressure as evaluated by clinical means
* Subjects with metal in the cranium
* Subjects with dental braces (but dental fillings are acceptable), metal fragments from occupational exposure or surgical clips in or near the brain

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44
Dates: Start 2006-05-05; Study Completion 2008-05-20

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Nutt JG, Muenter MD, Melton LJ 3rd, Aronson A, Kurland LT. Epidemiology of dystonia in Rochester, Minnesota. Adv Neurol. 1988;50:361-5. No abstract available. PMID 3400496